CLINICAL TRIAL: NCT00293865
Title: Prospective Multicentric Study of Sentinel Lymph Node Assessment Following Previous Surgical Biopsy for Early Breast Cancer
Brief Title: Study of Sentinel Lymph Node Assessment Following Previous Surgical Biopsy for Early Breast Cancer
Acronym: GATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 05/11-M
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast infiltrative cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: sentinel node — detection of the sentinel node in breast cancer
Procedure: GAS

SUMMARY:
The purpose of this study is to assess the detection rate and false negative rate of sentinel lymph node biopsy following previous surgical biopsy for early breast cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Previous conservative surgical biopsy
* Secondary pathological diagnosis of infiltrative cancer
* No clinically involved axillary node (N0)
* No previous neoadjuvant treatment
* Performance status European Cancer Conference (ECCO) Grade ≤ 1
* Patient's written informed consent to participate in the study according to French law
* Surgeon must have performed its learning curve

Exclusion Criteria:

* Lack of infiltrative breast carcinoma (in situ) pT4d > N0
* Breast cancer relapse
* Pregnancy
* Known patent blue allergy
* Indication for radical or partial mastectomy
* Patient unable to understand the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2006-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
false negatives

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Classe, MD, Principal Investigator — Centre Rene Gauducheau
Locations (17):
- France (17):
  - Hospîtal, Angers
  - Institut Bergonié, Bordeaux
  - Hospital, Brest
  - Centre Hospitalier, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - centre Léon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Alexis Vautrin, Nancy
  - Hospital, Nancy
  - Hopital Lariboisière, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Hospital, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre René Gauducheau, Saint-Herblain
  - Centre Claudius Regaud, Toulouse

REFERENCES:
- [Derived] Renaudeau C, Lefebvre-Lacoeuille C, Campion L, Dravet F, Descamps P, Ferron G, Houvenaeghel G, Giard S, Tunon de Lara C, Dupre PF, Fritel X, Ngo C, Verhaeghe JL, Faure C, Mezzadri M, Damey C, Classe JM. Evaluation of sentinel lymph node biopsy after previous breast surgery for breast cancer: GATA study. Breast. 2016 Aug;28:54-9. doi: 10.1016/j.breast.2016.04.006. Epub 2016 May 20. PMID 27214241